CLINICAL TRIAL: NCT06443619
Title: Efficacy of Glucose Addition to Bupivacaine in Serratus Anterior Plane Block to Reduce the Occurrence of Chronic Post-mastectomy Pain: A Randomized Controlled Trial
Brief Title: Efficacy of Glucose in Serratus Anterior Plane Block to Reduce the Occurrence of Chronic Post-mastectomy Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Alseoudy, Associate professor of Anesthesia, Intensive care and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.24.04.2582.
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Post-mastectomy Pain Syndrome
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): will receive unilateral USG-deep SAPB ; 15 ml 0.5 % isobaric bupivacaine with addition of 15ml glucose 10% to (30 ml total volume).
  Interventions: Procedure: unilateral USG-deep SAPB with glucose
- Group Π (Active Comparator): will receive unilateral USG-deep SAPB; 15ml 0.5% isobaric bupivacaine to be diluted with 15ml isotonic saline0.9% (30 ml total volume).
  Interventions: Procedure: unilateral USG-deep SAPB without glucose

INTERVENTIONS:
Procedure: unilateral USG-deep SAPB with glucose — patients will receive unilateral USG-deep SAPB ; 15 ml 0.5 % isobaric bupivacaine with addition of 15ml glucose 10% to (30 ml total volume).
  Arms: Group I
Procedure: unilateral USG-deep SAPB without glucose — will receive unilateral USG-deep SAPB; 15ml 0.5% isobaric bupivacaine to be diluted with 15ml isotonic saline0.9% (30 ml total volume).
  Arms: Group Π

SUMMARY:
Nearly 50% of patients suffer from chronic pain following breast cancer surgery. Several regional anesthesia techniques, including paravertebral block, erector spinae plane block, pectoral nerves block, and serratus anterior plane block, have been applied for acute pain control and prevention of chronic pain after breast cancer surgery. Exploiting the beneficial effect of glucose in regulating neuroinflammation and neuropathic pain, we hypothesize that the addition of glucose to bupivacaine could be superior to bupivacaine in ultrasound-guided SAPB in improving the quality of postoperative analgesia and preventing chronic pain after mastectomy. Patients will be randomly allocated into one of two equal groups (30 patients each ); the study group; Group I( B-D) (n=30): will receive unilateral USG-deep SAPB 0.4 ml/kg Of 0.25 % isobaric bupivacaine with addition of 15ml glucose 5% to (30 ml total volume); Group (B-N) (n=30): will receive unilateral USG-deep SAPB 0.4 ml/kg Of 0.25% isobaric bupivacaine to be diluted with 15ml isotonic saline (30 ml total volume). The occurence of postmastectomy pain, 3 months after surgery, will be the primary outcome.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed malignancy and the leading cause of cancer-related death in women. Although early detection and treatment have increased survival rates, chronic postsurgical pain (CPSP) is one of the most common complications of breast cancer surgery.

Nearly 50% of patients suffer from chronic pain following breast cancer surgery which is known as Post Mastectomy Pain Syndrome (PMPS). There are several risk factors for PMPS, including younger age, invasive surgical interventions, adjuvant radiation therapy following surgery, and high pain score in the early postoperative period. Several regional anesthesia (RA) techniques, including paravertebral block (PVB), pectoral nerves (PECS) block, and the erector spinae plane block (ESPB), have been applied for acute pain control and prevention of chronic pain after breast cancer surgery (BCS).

Recently, the serratus anterior plane block (SAPB) has become a newer interfacial plane block that appears to be safe and easily performed under ultrasound (de la Torre et al., 2014). A study concluded that preoperative SAPB with ropivacaine reduced the prevalence of CPSP at 3 months postoperativelyfrom 51.7% to 25.6%. Various adjuvants like fentanyl, clonidine, magnesium sulphate, nalbuphine, and dexamethasone have been used with bupivacaine in different blocks for prolonging the duration of analgesia and prevention of chronic pain. Using glucose 5% has been progressively applied to treat many peripheral entrapment neuropathies and has been proven to have outstanding effects in a few high-quality studies. Glucose 5% could decrease neurogenic inflammation by impeding the discharge of substance P and calcitonin gene-related peptides, which are pro-nociceptive substances that contribute to neurogenic inflammation and neuropathic pain. Exploiting the beneficial effect of glucose in regulating neuroinflammation and neuropathic pain, we hypothesize that the addition of glucose, as an adjuvant, to bupivacaine in the regional anesthesia technique for breast surgery could improve the quality of postoperative analgesia and prevent chronic pain after mastectomy. We hypothesize that the addition of glucose to bupivacaine could be superior to bupivacaine in ultrasound-guided SAPB in improving the quality of postoperative analgesia and preventing chronic pain after mastectomy. This randomized, double-blind study was designed to compare the efficacy and safety of co-administration of glucose and bupivacaine (study group), and bupivacaine alone (control group) in ultrasound-guided SAPB in patients undergoing modified radical mastectomy using the occurence of postmastectomy pain, 3 months after surgery, as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-II
* age ranging from 20 to 60 years
* scheduled for unilateral modified radical mastectomy

Exclusion Criteria:

* patient refusal to participate in the study
* infection at site of needle insertion
* hypersensitivity to the studied drugs
* psychotic disorders,
* bilateral MRM ,
* bleeding disorder
* chronic renal or hepatic diseases

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-06-04 (Estimated); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The prevalence of chronic pain (post mastectomy pain syndrome) | 3 months after surgery
  The prevalence of chronic pain (post mastectomy pain syndrome) of any severity: Numerical pain scale (NRS) >0 on a 0 - 10 scale

SECONDARY OUTCOMES:
Numerical pain scale (NRS) | over 24 hours
  Numerical pain scale (NRS) on a 0 - 10 scale, o no pain, 10 worst pain
Postoperative opioid consumption. | over 24 hours
  total consumption of morphine in the first 24 hours
Patient satisfaction with pain management | 24 hours
  Patient satisfaction with pain management assessed 24 h after surgery using an 11-point Likert scale (range, 0-10: 0, entirely unsatisfied; 10,fully satisfied).
The severity of CPSP and its impact on daily function | 3 and 6 months after surgery
  The severity of CPSP and its impact on daily function assessed 3 and 6 months after surgery using the revised brief pain inventory (BPI) Chinese-Simplified version